CLINICAL TRIAL: NCT00437645
Title: A Double-blind, Randomized, Multicenter, Parallel Group Study to Evaluate the Efficacy, Tolerability, and Safety of Treatment With the Combination of Valsartan/Amlodipine 160/5 mg Compared to Amlodipine 10 mg in Patients With Essential Hypertension Not Adequately Controlled With Amlodipine 5 mg Alone
Brief Title: Efficacy and Safety of Valsartan/Amlodipine Compared to Amlodipine in Patients With Essential Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Study Director, Novartis Pharmaceuticals
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CVAA489A2404
Record Dates: First submitted 2007-02-16; First posted 2007-02-21 (Estimated); Results first posted 2011-02-14 (Estimated); Last update posted 2014-11-11 (Estimated); Status verified 2014-11

CONDITIONS: Essential Hypertension
Keywords: Essential hypertension; blood pressure; edema; valsartan; amlodipine; combination treatment
MeSH Terms: conditions — Essential Hypertension; Edema | interventions — Valsartan; Amlodipine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Valsartan/amlodipine 160/5 mg (Experimental): Twelve (12) weeks treatment with the combination of valsartan/amlodipine 160/5 mg. Together with the active medication, patients received a placebo that matched amlodipine 5 mg. The three capsules were taken by mouth with water once daily in the morning, regardless of meals. Patients were instructed not to take their study medication the morning of their study visits. Instead, they brought the study medication with them to the site and took it there as instructed by the investigator.
  Interventions: Drug: Valsartan 160 mg capsules; Drug: Amlodipine 5 mg capsules; Drug: placebo
- Amlodipine 10 mg (Active Comparator): Eight (8) weeks of treatment with amlodipine 10 mg (two 5 mg capsules). Together with the active medication, the patients received a placebo that matched valsartan 160 mg. At Week 8, patients were switched and treated with the combination of valsartan/amlodipine 160/5 mg and a placebo that matched amlodipine 5 mg for an additional 4 weeks until the end of the study. The three capsules were taken by mouth with water once daily in the morning, regardless of meals. Patients were instructed not to take their study medication the morning of their study visits. Instead, they brought the study medication with them to the site and took it there as instructed by the investigator.
  Interventions: Drug: Valsartan 160 mg capsules; Drug: Amlodipine 5 mg capsules; Drug: placebo

INTERVENTIONS:
Drug: Valsartan 160 mg capsules
Drug: Amlodipine 5 mg capsules
Drug: placebo — capsules

SUMMARY:
This study was designed to compare the efficacy, tolerability, and safety of the combination valsartan/amlodipine 160/5 mg versus amlodipine 10 mg in patients with essential hypertension not adequately controlled (defined as mean sitting systolic blood pressure [msSBP] ≥ 130 mmHg and ≤ 160 mmHg) on amlodipine 5 mg alone. The study evaluated both the efficacy and tolerability of the treatments by providing data that assessed blood pressure and the proportion of patients developing peripheral edema.

ELIGIBILITY:
Inclusion Criteria:

* Male or female outpatients ≥ 55 years of age
* Patients with essential hypertension measured using a validated automated oscillometric device at Visit 1
* Non-treated patients must have a MSSBP ≥ 140 mmHg and ≤ 160 mmHg
* Patients pre-treated on monotherapy prior to Visit 1 must have MSSBP ≤ 160 mmHg
* To be eligible for randomization at Visit 2 (Day 1) all patients must have a MSSBP ≥ 130 mmHg and ≤ 160 mmHg
* No peripheral edema at Visit 2 (randomization)
* Written informed consent to participate in this study prior to any study procedures

Exclusion Criteria:

* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant
* Known or suspected contraindications, including history of allergy or hypersensitivity to angiotensin receptor blockers, calcium channel blockers, or to drugs with similar chemical structures
* Patients taking more than 1 antihypertensive medication at Visit 1
* Administration of any agent indicated for the treatment of hypertension after Visit 1 with the exception of pre-treated patients that require tapering down of anti-hypertensive treatments. For patients with previous antihypertensive medication that require a gradual downward titration, the tapering down should be done according to manufacturers instructions and last dose should be taken by week -2 prior to randomization
* msSBP > 180 mmHg or msDBP > 110 mmHg at any time between Visit 1 and Visit 2
* Evidence of a secondary form of hypertension, including but not limited to any of the following: Coarctation of the aorta, hyperaldosteronism, unilateral or bilateral renal artery stenosis, Cushing's disease, polycystic kidney disease, or pheochromocytoma
* History of hypertensive encephalopathy, cerebrovascular accident, transient ischemic attack, myocardial infarction, percutaneous coronary intervention (PCI) or coronary artery bypass graft surgery (CABG) 12 months prior to Visit 1
* History of heart failure Grade II - IV according to the NYHA classification
* Second or third degree heart block with or without a pacemaker
* Concomitant potentially life threatening arrhythmia or symptomatic arrhythmia
* Concomitant unstable angina pectoris
* Clinically significant valvular heart disease
* Patients with Type 1 diabetes mellitus
* Patients with Type 2 diabetes mellitus who are not well controlled based on the investigator's judgment. It is recommended that Type 2 diabetic patients are adequately controlled and, if treated with medication, be on a stable dose of oral anti-diabetic medication for at least 4 weeks prior to Visit 1
* Evidence of hepatic disease as determined by one of the following: AST or ALT values > 2x UNL at study entry, a history of hepatic encephalopathy, history of esophageal varices, or history of portocaval shunt
* Evidence of renal impairment as determined by one of the following: serum creatinine > 1.5 x UNL at visit 1, history of dialysis, or history of nephrotic syndrome
* Serum potassium values > 5.5 mmol/L at study entry
* Any surgical or medical condition which might significantly alter the absorption, distribution, metabolism or excretion of any drug
* Any surgical or medical condition which, at the discretion of the investigator or Novartis medical monitor, places the patient at higher risk from his/her participation in the study, or is likely to prevent the patient from complying with the requirements of the study or completing the study period
* Volume depletion based on the investigator's clinical judgment using vital signs, skin turgor, moistness of mucous membranes, and laboratory values
* Any severe, life-threatening disease within the past five years
* History of drug or alcohol abuse within the last 2 years
* Use of other investigational drugs at the time of enrollment, or within 30 days or 5 half-lives of enrollment, whichever is longer
* Inability to communicate and comply with all study requirements including the unwillingness or inability to provide informed consent
* Persons directly involved in the execution of this protocol

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1183 (Actual)
Dates: Start 2007-01; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Chair — Novartis Pharmaceuticals
Locations (12):
- sites in Argentina, Agentina, Argentina
- sites in Chile, Chile, Chile
- sites in Ecuador, Ecuador, Ecuador
- sites in Finland, Finland, Finland
- sites in France, France, France
- sites in Germany, Germany, Germany
- sites in Italy, Italy, Italy
- sites in Norway, Norway, Norway
- sites in Spain, Spain, Spain
- sites in Sweden, Sweden, Sweden
- sites in Switzerland, Switzerland, Switzerland
- sites in Turkey, Turkey, Turkey (Türkiye)

REFERENCES:
- [Derived] Schrader J, Salvetti A, Calvo C, Akpinar E, Keeling L, Weisskopf M, Brunel P. The combination of amlodipine/valsartan 5/160 mg produces less peripheral oedema than amlodipine 10 mg in hypertensive patients not adequately controlled with amlodipine 5 mg. Int J Clin Pract. 2009 Feb;63(2):217-25. doi: 10.1111/j.1742-1241.2008.01977.x. PMID 19196360

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Valsartan/Amlodipine 160/5 mg | Amlodipine 10 mg
Started | 592 | 591
Completed | 557 | 476
Not Completed | 35 | 115
Not completed — Adverse Event | 15 | 84
Not completed — Withdrawal by Subject | 10 | 22
Not completed — Protocol Violation | 3 | 3
Not completed — Lost to Follow-up | 2 | 3
Not completed — Administrative problems | 2 | 1
Not completed — Lack of Efficacy | 2 | 1
Not completed — Condition no longer requires study drug | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Valsartan/Amlodipine 160/5 mg | Amlodipine 10 mg | Total
Number analyzed (Participants) | 592 | 591 | 1183
Age, Continuous [Mean (Standard Deviation); unit: Age (years)]
  Overall study | 65.6 (7.56) | 65.4 (7.16) | 65.5 (7.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 285 | 284 | 569
  Male | 307 | 307 | 614

OUTCOME MEASURES:

1. Primary Outcome: Change in Mean Sitting Systolic Blood Pressure (msSBP) From Baseline to Week 8
Description: Blood pressure (BP) was measured at trough (24±3 hours post-dose). The arm in which the highest sitting diastolic BP was found at study entry was used for all subsequent readings. If there was < 0. 5 mmHg difference in BP between the 2 arms, the non-dominant arm was used. At each visit, after the patient was in a sitting position with the back supported and both feet placed on the floor for 5 minutes, systolic and diastolic BP were measured 3 times with an automated BP monitor and appropriate size cuff. Means of the 3 measurements were calculated. A negative change indicates lowered BP.
Time Frame: Baseline to Week 8
Population: Intent-to-treat (ITT) population: All randomized patients who had a baseline and at least one post-baseline efficacy assessment. For patients who discontinued prior to Week 8, the last post-baseline msSBP measurement collected was used for the analysis (last observation carried forward [LOCF]).
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Valsartan/Amlodipine 160/5 mg | Amlodipine 10 mg
Number analyzed (Participants) | 567 | 510
mmHg | -8.01 (0.5944) | -6.30 (0.6088)
Statistical Analysis 1: Comparison: Valsartan/Amlodipine 160/5 mg vs Amlodipine 10 mg; Test type: Non-Inferiority or Equivalence — Statistical analysis for non-inferiority of valsartan/amlodipine 160/5 mg to amlodipine 10 mg alone with a non-inferiority margin of 3 mm Hg; ANCOVA; Mean Difference (Final Values) = -1.72, 95% CI 2-sided [-3.00 to -0.44], Standard Error of Mean 0.65

2. Primary Outcome: Percentage of Patients With Peripheral Edema From Baseline to Week 8
Description: Only occurrences of peripheral edema quantified as a reported adverse event coded as peripheral edema were included in the analysis. If a patient experienced more than one occurrence of peripheral edema between Day 1 and Week 8, it was only counted once in the analysis.
Time Frame: Baseline to Week 8
Population: Safety population: All randomized patients.
Measure: Number; unit: Percentage of patients
Arm/Group | Valsartan/Amlodipine 160/5 mg | Amlodipine 10 mg
Number analyzed (Participants) | 592 | 591
Percentage of patients | 6.6 | 31.1

3. Secondary Outcome: Change in Mean Sitting Diastolic Blood Pressure (msDBP) From Baseline to Week 8
Description: as for outcome 1
Time Frame: Baseline to Week 8
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Valsartan/Amlodipine 160/5 mg | Amlodipine 10 mg
Number analyzed (Participants) | 567 | 510
mmHg | -4.65 (0.3616) | -4.13 (0.3690)

4. Secondary Outcome: Change in Mean Sitting Systolic and Diastolic Blood Pressure (msSBP, msDBP) From Baseline to Weeks 4, 8, and 12
Description: as for outcome 1
Time Frame: Baseline to Weeks 4, 8, and 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Valsartan/Amlodipine 160/5 mg | Amlodipine 10 mg
Number analyzed (Participants) | 576 | 535
mmHg
  msSBP: Week 4 (n=576, 535) | -8.40 (0.5559) | -6.48 (0.5676)
  msSBP: Week 8 (n=567, 510) | -8.15 (0.6065) | -6.11 (0.6266)
  msSBP: Week 12 (n=569, 531) | -9.08 (0.6968) | -7.82 (0.7088)
  msDBP: Week 4 (n=576, 535) | -5.05 (0.3559) | -4.23 (0.3623)
  msDBP: Week 8 (n=576, 510) | -4.68 (0.3632) | -3.97 (0.3736)
  msDBP: Week 12 (n=569, 531) | -5.50 (0.03735) | -4.90 (0.3785)

5. Secondary Outcome: Percentage of Patients Achieving a Systolic Response at Weeks 4, 8, and 12
Description: Systolic response was defined as msSBP < 130 mmHg or at least a 20 mmHg reduction from baseline in msSBP at Weeks 4, 8, and 12. Blood pressure (BP) was measured at trough (24±3 hours post-dose). The arm in which the highest sitting diastolic BP was found at study entry was used for all subsequent readings. At each visit, after the patient was in a sitting position with the back supported and both feet placed on the floor for 5 minutes, systolic and diastolic BP were measured 3 times with an automated BP monitor and appropriate size cuff. Means of the 3 measurements were calculated.
Time Frame: Baseline to Weeks 4, 8, and 12
Population: as for outcome 1
Measure: Number; unit: Percentage of patients
Arm/Group | Valsartan/Amlodipine 160/5 mg | Amlodipine 10 mg
Number analyzed (Participants) | 576 | 535
Percentage of patients
  Week 4 (n=576, 535) | 35.07 | 25.42
  Week 8 (n=567, 510) | 34.22 | 25.49
  Week 12 (n=569, 531) | 37.96 | 31.26

ADVERSE EVENTS:
Arm/Group | Valsartan/Amlodipine 160/5 mg | Amlodipine 10 mg
Serious Adverse Events (participants affected / at risk) | 11/592 | 8/591
Other Adverse Events (participants affected / at risk) | 61/592 | 201/591
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Valsartan/Amlodipine 160/5 mg (N=592) | Amlodipine 10 mg (N=591)
Atrial fibrillation (Cardiac disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastrointestinal necrosis (Gastrointestinal disorders) | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 1
Asthenia (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 2 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Hantavirus pulmonary infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Drug toxicity (Injury, poisoning and procedural complications) | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1
Ligament rupture (Injury, poisoning and procedural complications) | 1 | 0
Meniscus lesion (Injury, poisoning and procedural complications) | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Dysphasia (Nervous system disorders) | 0 | 1
Neglect of personal appearance (Psychiatric disorders) | 0 | 1
Bladder tamponade (Renal and urinary disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 0
Renal impairment (Renal and urinary disorders) | 1 | 0
Epididymitis (Reproductive system and breast disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Valsartan/Amlodipine 160/5 mg (N=592) | Amlodipine 10 mg (N=591)
Oedema peripheral (General disorders) | 43 | 186
Headache (Nervous system disorders) | 18 | 33

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Disclosure Restriction Description: The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.